CLINICAL TRIAL: NCT06777368
Title: REdo tranScatheter Aortic Valve Replacement for Transcatheter aOrtic Valve failuRE
Acronym: RESTORE
Status: Recruiting | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT23040EVR015
Record Dates: First submitted 2024-12-17; First posted 2025-01-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Medtronic Transcatheter Aortic Valves (TAV) or Edwards Transcatheter Aortic Valves (TAV): Subjects will receive either a Medtronic TAV or Edwards TAV
  Interventions: Device: Medtronic TAV; Device: Edwards TAV

INTERVENTIONS:
Device: Medtronic TAV — Medtronic TAV where commercially available
Device: Edwards TAV — Edwards TAV where commercially available.

SUMMARY:
The purpose of this study is to generate clinical evidence on valve safety and performance in subjects treated by redo Transcatheter Aortic Valve Replacement (TAVR).

DETAILED DESCRIPTION:
Primary Objectives:

* To determine the acute and long-term outcomes of redo TAVR for the treatment of BVF affecting TAVs
* To determine the factors which are associated with the acute and long-term outcomes of redo TAVR

ELIGIBILITY:
Inclusion Criteria:

* BVF of a TAV (either Medtronic or Edwards) requiring redo TAVR

Exclusion Criteria:

* BVF due solely to paravalvular regurgitation
* Active endocarditis
* Untreated acute valve thrombosis
* Life-expectancy less than 1-year
* Subject is less than legal age of consent, legally incompetent, or otherwise vulnerable
* Participating in another study that may influence the outcome of this study

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with symptomatic heart disease due to BVF affecting TAVs and requiring redo TAVR.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | Early (30-days)
  30-day redo TAVR success defined as correct positioning of a single redo prosthetic heart valve into the proper anatomic location, intended performance of the valve (mean gradient <20mmHg, peak velocity <3 m/s, Doppler velocity index (DVI) ≥0.25, aortic regurgitation (AR) < moderate), and freedom from all-cause mortality, coronary obstruction, unplanned coronary revascularization, and surgery or intervention related to the device
Primary Outcome Measure | Late (1-year)
  a composite endpoint of 1-year freedom from all-cause mortality, all stroke, or any re-hospitalization for valve or redo TAVR procedure-related causes

SECONDARY OUTCOMES:
Valve Academic Research Consortium (VARC) 3 technical success (at exit from procedure room) | Time of procedure
  (VARC) 3 technical success (at exit from procedure room)
VARC 3 30-day device success | 30-Day
  30-day device success
VARC 3 30-day early safety | 30-Day
  30-day early safety
Peak and mean invasive gradient post-procedure | Time of procedure
  Peak and mean invasive gradient will be measured in mmHg
In-hospital clinical outcomes | Treatment up to 7 days (or until patient is discharged from the hospital if later than 7 days)
  Percentage of all participants with all-cause mortality, all stroke, Myocardial infarction (MI), Coronary artery obstruction, Unplanned Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Grafting (CABG), Bleeding (VARC 3 type 1-4), Major and Minor vascular and access-related complications, Cardiac structural complications, Permanent pacemaker implantation (PPI), Acute Kidney Injury (AKI) stage 1-4, Endocarditis, and Valve Thrombosis.
Clinical outcomes at 30 days, 1-year, and annually thereafter | 30 days, at 1 year, at 2 years, at 3 years, at 4 years, and at 5 years.
  All-cause mortality, All stroke, Myocardial infarction (MI), Coronary artery obstruction, Bleeding (VARC 3 type 1-4), Major and Minor vascular and access-related complications, Cardiac structural complications, Permanent pacemaker implantation (PPI), Acute Kidney Injury (AKI) stage 1-4, Endocarditis, Valve Thrombosis, Any rehospitalization and re-intervention.
Bioprosthetic Valve Dysfunction (BVD) at the final required follow-up visit | 5 year
  Intrinsic permanent changes to the prosthetic valve, including wear and tear, leaflet disruption, flail leaflet, leaflet fibrosis and/or calcification, or strut fracture or deformation
Bioprosthetic Valve Failure (BVF) at the final required follow-up visit | Through study completion or Up to 5-years
  Any bioprosthetic valve dysfunction associated with clinically expressive criteria (new-onset or worsening symptoms, left ventricle dilation/hypertrophy/dysfunction, or pulmonary hypertension) or irreversible Stage 3 Hemodynamic Valve Deterioration (HVD) or Aortic valve reoperation or re-intervention, or Valve-related death.
Echocardiographic assessment pre-discharge or at 30 days, 1-year, and annually thereafter | After the procedure and prior to discharge from the hospital, at 30 days, at 1 year, at 2 years, at 3 years, at 4 years, and at 5 years.
  Left ventricular ejection fraction, mean gradient across aortic valve, effective orifice area, effective orifice area index, patient-prosthesis mismatch, Doppler Velocity Index, total aortic regurgitation, paravalvular aortic regurgitation, and transvalvular aortic regurgitation.
Evaluate coronary accessibility (e.g., commissural alignment, valve to valve alignment, etc.) based on Computed Tomography (CT) at either pre-discharge or 30 days | Up to 30 days
  Evaluate coronary accessibility
New York Heart Association (NYHA) classification at pre-discharge, 30 days, 1-year, and annually thereafter | After the procedure and prior to discharge from the hospital, at 30 days, at 1 year, at 2 years, at 3 years, at 4 years, and at 5 years.
  New York Heart Association (NYHA) classification
KCCQ Quality of life (QoL) assessments at 30 days, 1-year, and annually thereafter | At 30 days, at 1 year, at 2 years, at 3 years, at 4 years, and at 5 years.
  QoL: KCCQ assessment
EQ5D Quality of life (QoL) assessments at 30 days, 1-year, and annually thereafter | At 30 days, at 1 year, at 2 years, at 3 years, at 4 years, and at 5 years.
  QoL: EQ5D assessment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Fontana, MD, Study Chair — Los Robles Regional Medical Center; Guilherme Attizzani, MD, Principal Investigator — UH, Cleveland Medical Center; Basel Ramlawi, Principal Investigator — Lankenau Heart Institute
Locations (70):
- United States (70):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Sutter Heatlh, Sacramento, California
  - Kaiser Permanente Northern California, Sacramento, California
  - Stanford Hospital & Clinics, Stanford, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Medical Center of the Rockies, Loveland, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - MedStar Washington Medical Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - HealthPark Medical Center, Lee Memorial Health, Fort Myers, Florida
  - Orlando Health/Orlando Regional Medical Center, Orlando, Florida
  - Tampa General/USF, Tampa, Florida
  - Parkview Health, Fort Wayne, Indiana
  - Saint Vincent Heart Center of Indiana, Indianapolis, Indiana
  - MercyOne Iowa Heart Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - The University of Kansas, Kansas City, Kansas
  - Ascension Via Christi St. Francis, Wichita, Kansas
  - Maine Medical Center, Portland, Maine
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health (Spectrum), Grand Rapids, Michigan
  - Abbott Northwestern/Minneapolis Heart, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Providence Saint Patrick Hospital, Missoula, Montana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Saint Francis Hospital, Roslyn, New York
  - Montefiore Medical Center, The Bronx, New York
  - Astrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland Medical Center, Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - UPMC Pinnacle, Mechanicsburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - St. Thomas West Hospital, Nashville, Tennessee
  - Ascension Seton Medical Center Austin, Austin, Texas
  - Heart Hospital of Austin, Austin, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Providence Heart Institute (Providence Sacred Heart), Spokane, Washington
  - Aurora St. Lukes Medical Center, Milwaukee, Wisconsin
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No